CLINICAL TRIAL: NCT05257629
Title: Aggressive Smoking Cessation Therapy Among People at Elevated Cardiovascular Risk (ASAP) Trial
Brief Title: Aggressive Smoking Cessation Trial (ASAP)
Acronym: ASAP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Mark Eisenberg, MD, Principal Investigator, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ASAP-001, Version 10
Record Dates: First submitted 2022-02-01; First posted 2022-02-25 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Acute Coronary Syndrome; Cardiovascular Diseases
Keywords: acute coronary syndrome; smoking cessation; randomized controlled trial; varenicline; e-cigarettes; cardiovascular disease
MeSH Terms: conditions — Acute Coronary Syndrome; Cardiovascular Diseases; Smoking Cessation; Vaping | interventions — Varenicline; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination Therapy Arm (Varenicline and Nicotine E-Cigarettes Plus Counseling) (Active Comparator): Patients in the combination therapy arm will be supplied funds and instructions for the purchase of e-cigarettes and cartridges/pods upon hospital discharge and at the week 4 and 12 clinic visits. As with standard NRTs such as the gum, inhaler, and lozenge, the investigators expect smokers will self-regulate administration according to their withdrawal symptoms. Use will be monitored via self-report for telephone follow-ups. At clinic visits, patients will be asked to bring their e-cigarettes, used and unused cartridges/pods, and purchasing receipts. Patients will be advised regarding the signs and symptoms of nicotine toxicity and of an allergic reaction.
  Interventions: Combination Product: Combination Therapy Arm (Varenicline and Nicotine E-Cigarettes Plus Counseling)
- Varenicline Plus Counseling (Other): All patients will begin varenicline in-hospital upon randomization. For the first 3 days, patients will take a 0.5 mg tablet once a day. They will then take a 0.5 mg tablet twice a day for the following 4 days, and one 1 mg tablet twice a day from day 8 onward for the remainder of the 12-week treatment. Use will be monitored via self-report for telephone follow-ups and return of all unused tablets at the end of the treatment period. Should a patient experience severe side effects (such as headache, nausea, vomiting, dizziness, dyspepsia, fatigue, insomnia, abnormal dreams, constipation, or flatulence) on day 8 onward, the varenicline dose should be reduced from 1 mg twice daily to 0.5 mg twice daily prior to study medication discontinuation.
  Interventions: Other: Varenicline Plus Counseling

INTERVENTIONS:
Combination Product: Combination Therapy Arm (Varenicline and Nicotine E-Cigarettes Plus Counseling) — Varenicline and nicotine e-cigarettes plus counseling
  Arms: Combination Therapy Arm (Varenicline and Nicotine E-Cigarettes Plus Counseling)
Other: Varenicline Plus Counseling — Varenicline plus counseling
  Arms: Varenicline Plus Counseling

SUMMARY:
The ASAP Trial is a 5-year, multi-centre, randomized controlled trial that will assess the efficacy, safety, and tolerability of aggressive smoking cessation therapy among people at elevated cardiovascular risk. It will recruit 798 adult patients smoking on average at least 10 conventional (tobacco) cigarettes per day who are motivated to quit smoking and have either been diagnosed with ACS requiring hospitalization or are outpatients at elevated cardiovascular risk. Patients will be randomized (1:1) to one of two treatment arms: (1) combination therapy of varenicline and nicotine e-cigarettes plus counseling or (2) varenicline plus counseling for 12 weeks, with 52-week follow-up.

DETAILED DESCRIPTION:
Background and Importance:

People who smoke are at an elevated risk of developing cardiovascular disease (CVD). Those who have an acute coronary syndrome (ACS), including myocardial infarction and unstable angina, and continue to smoke have a 35% increased risk of reinfarction or death compared with those who quit. Our previous smoking cessation trials have established varenicline (Champix) as the "gold standard" for patients with CVD. However, more than 50% of patients motivated to quit who receive varenicline for 12 weeks immediately post-ACS will return to smoking within 6 months. Therefore, more effective smoking cessation strategies are needed. Based on newly available data from randomized controlled trials (RCTs), including our E3 Trial, which suggest that nicotine e-cigarettes are more efficacious for smoking cessation than other nicotine replacement therapies and counseling alone, the investigators propose to combine varenicline and nicotine e-cigarettes (aggressive smoking cessation therapy). The proposed aggressive therapy is a novel approach needed now to increase abstinence in people at elevated cardiovascular risk.

Goal(s)/Research Aims:

The Aggressive Smoking Cessation Therapy Among People at Elevated Cardiovascular Risk (ASAP) Trial is a 5-year, multi-centre RCT that will assess the efficacy, safety, and tolerability of aggressive smoking cessation therapy among people at elevated cardiovascular risk. The specific aims are:

1. To assess the efficacy of combination therapy (varenicline and nicotine e-cigarettes) versus varenicline alone for 12 weeks, in terms of biochemically-validated 7-day point prevalence and continuous smoking abstinence, and ≥50% reduction in daily cigarette consumption at 24 and 52 weeks among people at elevated cardiovascular risk.
2. To describe the safety and tolerability of varenicline combined with nicotine e-cigarettes, in terms of serious adverse events (SAEs), adverse events (AEs), treatment discontinuation due to side effects, and therapy adherence over the 12-week treatment period.

Methods/Approaches/Expertise:

A total of 798 participants will be randomized 1:1 to: (1) varenicline and nicotine e-cigarettes (aggressive smoking cessation therapy), or (2) varenicline alone for 12 weeks, with follow-up of 52 weeks. Both arms will receive individual smoking cessation counseling. Participants randomized to aggressive therapy (varenicline and nicotine e-cigarette) will be given funds to cover the purchase of e-cigarettes and nicotine cartridges. Funds will be provided at baseline for the first 4 weeks of e-cigarette use. Participants who follow the e-cigarette purchasing instructions and provide receipts at subsequent clinic visits will be provided additional funds at week 4 (for weeks 4 to 8) and reimbursed at week 12 (for weeks 8 to 12). Participants will begin varenicline (titrated to 1.0 mg twice daily) and counseling at baseline, and e-cigarette use (if applicable) after the baseline visit. Eligible people will have or be at elevated risk of developing CVD, self-identify as regular smokers (≥10 cigarettes/day for ≥1 year), and be motivated to quit. They will complete telephone follow-ups at weeks 1, 2, 8, and 18, and clinic visits at weeks 4, 12, 24, and 52. We will collect information about self-reported smoking, treatment adherence, and adverse events. Self-reported smoking abstinence will be biochemically-validated at clinic visits using exhaled carbon monoxide (≤10 ppm). The primary endpoint will be biochemically-validated 7-day point prevalence smoking abstinence at 24 weeks. With 399 participants per arm and an alpha of .05, the investigators will have 80% power to detect a ≥10% difference in abstinence at 24 weeks. The ASAP Trial will be conducted by a highly experienced team of researchers and enrolling centres, who have previously completed three smoking cessation RCTs, including two in cardiac patients.

Expected Outcomes:

Smoking cessation is essential to reduce morbidity and mortality in this high-risk patient population. ASAP will provide regulators, health care professionals, and smokers with important information about the efficacy of aggressive varenicline and nicotine e-cigarettes therapy for smoking cessation in people at an elevated cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

1. Patients currently hospitalized or being discharged from hospital who have suffered an ACS, defined as follows:

   i. MI, defined by positive troponin T, troponin I, or CK-MB levels (as defined by institution-specific cut-offs) and ≥ 1 of the following:
   1. Ischemic symptoms for ≥ 20 min;
   2. Electrocardiogram (ECG) changes indicative of ischemia (ST-segment elevation or depression);
   3. Development of pathological Q waves on the ECG

   ii. Unstable angina with significant coronary artery disease, defined by all of the following:
   1. Ischemic symptoms for ≥ 20 min;
   2. ECG changes indicative of ischemia (ST-segment changes);
   3. At least one lesion ≥ 50% on angiogram performed during the current hospitalization.

   [Note: patients who undergo cardiac catheterization or percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) surgery will be eligible provided they are able to start varenicline in-hospital and nicotine e-cigarette at discharge.]

   OR

   Outpatients with the following diagnoses/conditions:

   i. Cardiovascular:
   1. Coronary artery disease documented with angiography or coronary CT;
   2. Previous ACS, MI, stable or UA;
   3. Previous coronary revascularization (e.g. PCI or CABG). ii. Renovascular:

   a. Chronic kidney disease. iii. Cerebrovascular:

   a. Previous cerebral infarction or transient cerebral ischemic attack. iv. Peripheral vascular:
   1. Abdominal aortic aneurysm > 3.0 cm or previous aortic aneurysm surgery;
   2. Ankle-brachial pressure index of < 0.9 or intermittent claudication;
   3. Documented carotid artery disease;
   4. Lower-limb amputation;
   5. Previous lower-limb bypass surgery or angioplasty.

   v. ≥1 risk factors:
   1. BMI ≥ 27 kg/m2;
   2. Dyslipidemia;
   3. Family history (first degree relative: parents or siblings only) of coronary heart disease or stroke before the age of 60 years;
   4. Hypertension;
   5. Males aged ≥ 55 years/females aged ≥ 60 years;
   6. Diabetes mellitus. vi. Heart-related conditions:

   <!-- -->

   1. Atrial fibrillation or flutter;
   2. Cardiomyopathy;
   3. Heart failure;
   4. Left ventricular hypertrophy (evidenced by echocardiography or ECG);
   5. Valvular disease (evidenced by echocardiography).
2. Smoked on average ≥ conventional cigarettes/day for the past year;
3. Age ≥18 years;
4. Motivated to quit smoking according to the Motivation To Stop Scale (MTSS) (≥ level 5);
5. Able to understand and provide informed consent in English or French;
6. If randomized to the combination arm (varenicline and e-cigarette plus counseling), willing and able to purchase e-cigarettes with the following properties: rechargeable, closed system that uses sealed cartridges or pods, tobacco or no flavor only, and nicotine strength of 20 mg/ml (2%) or less;
7. Likely to be available for 52 weeks of follow-up.

Exclusion Criteria:

1. Pregnant or lactating females;
2. Use of any of the following in the 30 days prior to eligibility assessment:

   i. Varenicline or bupropion for smoking cessation; ii. Nicotine or non-nicotine e-cigarettes; iii. Other anti-craving medication (e.g., naltrexone, acamprosate) with the potential to alter substance-seeking behaviors;
3. Use of nicotine replacement therapy (NRT) in the 7 days prior to eligibility assessment [Note: If participant is prescribed non-study NRT while hospitalized, they can continue using the non-study NRT until being discharged, even while taking the investigational products. Upon discharge, use of the non-study NRT should be stopped.];
4. Use of varenicline or e-cigarettes (nicotine or non-nicotine) for ≥14 days consecutively in the past year;
5. Previous serious adverse reaction to varenicline and/or e-cigarettes (nicotine or non-nicotine);
6. NYHA or Killip Class III or IV at the time of randomization;
7. Any unstable psychiatric disorder (as per enrolling physician);
8. Renal impairment with creatinine levels ≥2 times upper limit of normal or eGFR ≤15;
9. Use of any illegal drugs in the past year;
10. Planned use of cannabis (smoked) or other tobacco products (smoked or other) during the study period. [Note: use of cannabis which is not smoked is permitted (e.g., edibles, ingested or vaped oils). However, methods which involve combustion could invalidate biochemical validation via exhaled carbon monoxide.]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 798 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2026-03-07 (Estimated); Study Completion 2027-03-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with 7-day point prevalence smoking abstinence | 24 weeks
  Biochemically-validated 7-day point prevalence smoking abstinence at 24 weeks, defined as self-reported abstinence in the past 7 days with exhaled carbon monoxide ≤ 10 ppm.

SECONDARY OUTCOMES:
Number of participants with continuous smoking abstinence | 1, 2, 8, and 18 weeks
  Biochemically-validated continuous abstinence at 4, 12, and 24 weeks, defined as self-reported abstinence since baseline with exhaled carbon monoxide ≤ 10 ppm at all clinic follow-ups, and self-reported 0 cigarette smoked in the past 7 days at telephone follow-ups (1, 2, 8, and 18 weeks).
Number of participants with prolonged smoking abstinence | 4, 8, 12, 18, and 24 weeks
  Prolonged abstinence, defined as self-reported abstinence at all clinical and telephone follow-ups after an initial 2-week grace period with exhaled carbon monoxide ≤ 10 ppm at 4, 12, and 24 weeks, and self-reported 0 cigarette smoked in the past 7 days at the 8, and 18 weeks telephone follow-ups.
Change in daily cigarette consumption | 24 weeks
  Change in self-reported daily conventional cigarette consumption from baseline compared to 24 weeks.
Number of participants with ≥50% reduction in daily cigarette consumption | 24 weeks
  Proportion of participants with ≥50% reduction in self-reported daily cigarette consumption from baseline compared to 24-weeks.
Number of participants with point prevalent abstinence or ≥50% reduction in daily cigarette consumption at 24 weeks | 24 weeks
  Composite endpoint of point prevalent abstinence or ≥50% reduction in daily cigarette consumption at 24 weeks
Frequency of Serious Adverse Events (SAEs) | 12 weeks
  The number of serious adverse events (SAE) reported over the 12 week treatment period.
  A SAE is defined as an adverse event which requires in-patient hospitalization or prolongation of existing hospitalization, that causes congenital malformation, that results in persistent or significant disability or incapacity, that is life-threatening, or that results in death.
Frequency of Adverse Events (AEs) | 12 weeks
  The number of adverse events reported over the 12 week treatment period. An adverse event is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of the trial drug, whether or not considered related to the e-cigarettes or varenicline.
Frequency of drop-outs | 12 weeks
  The number of drop-outs due to side effects of the e-cigarettes or varenicline over the 12 week treatment period.
Spirometry measurements (subset) | 24 weeks
  For a sub-set of 100 patients, 50 from each arm, randomized at 4-5 recruiting sites, undergoing spirometry measurements, differences in FVC, FEV1, and FEV1/FVC ratio as well as measures of small airways disease between pre- and post-bronchodilator at week 24 from baseline.
O2 Cost Diagram and COPD Assessment Test (subset) | 24 weeks
  For the same sub-set of 100 patients undergoing spirometry measurements randomized at 4-5 recruiting sites, the difference in the O2 Cost Diagram and the CAT at week 24 from baseline.

OTHER OUTCOMES:
Number of patients with 7-day point prevalence smoking abstinence at 4, 12, and 52 weeks | 4, 12, and 52 weeks
  Biochemically-validated 7-day point prevalence smoking abstinence at 4, 12, and 52 weeks, defined as self-reported abstinence in the past 7 days with exhaled carbon monoxide ≤ 10 ppm.
Number of patients with continuous abstinence at 4, 12, 24, and 52 weeks | 4, 12, 24, and 52 weeks
  Biochemically-validated continuous abstinence at 4, 12, 24, and 52 weeks, defined as self-reported abstinence since baseline with exhaled carbon monoxide ≤ 10 ppm at all follow-up visits.
Number of prolonged smoking abstinence at all follow-up visits | 4, 12, 24, and 52 weeks
  Prolonged abstinence, defined as self-reported abstinence at all follow-up visits after an initial 2 weeks grace period with exhaled carbon monoxide ≤ 10 ppm at 4, 12, 24, and 52 weeks.
Change in daily cigarette consumption at all other weeks | 1, 2, 4, 8, 12, 18, and 52 weeks
  Change in self-reported daily conventional cigarette consumption from baseline at weeks 1, 2, 4, 8, 12, 18, and 52.
Number of patients with ≥50% reduction in daily cigarette consumption at all other weeks | 1, 2, 4, 8, 12, 18, and 52 weeks
  Proportion of participants with ≥50% reduction in self-reported daily cigarette consumption from baseline at weeks 1, 2, 4, 8, 12, 18, and 52.
Number of participants with point prevalent abstinence or ≥50% reduction in daily cigarette consumption at all other weeks | 1, 2, 4, 8, 12, 18, and 52 weeks
  Composite endpoint of point prevalent abstinence or ≥50% reduction daily cigarette consumption at weeks 1, 2, 4, 8, 12, 18, and 52.
Spirometry measurements (subset) at all other clinic visits | 4, 12, and 52 weeks
  For the sub-set of 100 patients undergoing spirometry measurements, differences in FVC, FEV1, and FEV1/FVC ratio as well as measures of small airways disease between pre- and post-bronchodilator at week 4, week 12, and week 52.
O2 Cost Diagram and COPD Assessment Test (subset) at all other clinic visits | 4, 12, and 52 weeks
  For the sub-set of 100 patients undergoing spirometry measurements, the difference in the O2 Cost Diagram and the CAT at weeks 4, 12, and 52 compared to baseline.
Number of patients averaging ≥1 pill of varenicline/day | 12 weeks
  To describe the proportion of participants averaging ≥1 pill/day for varenicline over the treatment period.
To describe e-cigarette pattern of use | 12 weeks
  To describe the nicotine e-cigarette pattern of use during the treatment period in terms of self-reported average sessions per week, and puffs per session (7-day recall).

CONTACTS AND LOCATIONS:
Locations (13):
- Canada (13):
  - Fraser Clinical Trials, New Westminster, British Columbia
  - Dr. Georges-L.-Dumont University Hospital Center, Moncton, New Brunswick
  - NL Health Sciences, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - St. Joseph's Hospital, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Hospitalier de L'Universite de Montreal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No